CLINICAL TRIAL: NCT03719664
Title: A Phase 2, Multicenter, Three-part Study to Establish the Dosage, Safety and Antiviral Activity of Combination Therapy With Albuvirtide and 3BNC117 as Long-Acting Maintenance Therapy in Virologically Suppressed Subjects With HIV-1 Infection
Brief Title: Albuvirtide and 3BNC117 as Long-Acting Maintenance Therapy in Virologically Suppressed Subjects
Acronym: ABL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Frontier Biotechnologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABT-3BNC117_201
Record Dates: First submitted 2018-10-22; First posted 2018-10-25 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: HIV-1-infection
Keywords: HIV-1; 3BNC117; Albuvirtide; Broadly neutralizing antibody; Long-Acting HIV-1 Fusion Inhibitor
MeSH Terms: interventions — albuvirtide; HIV Fusion Inhibitors; 3BNC117 antibody; Antibodies, Monoclonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1: albuvirtide & 3BNC117 (Experimental): albuvirtide 0.32 g and 3BNC117 2 g every 2 weeks
  Interventions: Drug: Albuvirtide; Drug: 3BNC117
- Cohort 2: albuvirtide & 3BNC117 (Experimental): albuvirtide 0.32 g and 3BNC117 2 g every 4 weeks
  Interventions: Drug: Albuvirtide; Drug: 3BNC117
- Control Arm 1: Baseline ART (Active Comparator): Subjects continuing on baseline ART
  Interventions: Drug: Baseline ART
- Cohort 3: albuvirtide & 3BNC117 (Experimental): albuvirtide 0.32 g and 3BNC117 0.8 g every 4 weeks
  Interventions: Drug: Albuvirtide; Drug: 3BNC117
- Cohort 4: albuvirtide & 3BNC117 (Experimental): albuvirtide 0.16 g and 3BNC117 0.8 g every 4 weeks
  Interventions: Drug: Albuvirtide; Drug: 3BNC117
- Optimal Dose: albuvirtide & 3BNC117 (Experimental): albuvirtide and 3BNC117 every 2 or 4 weeks
  Interventions: Drug: Albuvirtide; Drug: 3BNC117
- Control Arm 2: Baseline ART (Active Comparator): Subjects continuing on baseline ART
  Interventions: Drug: Baseline ART

INTERVENTIONS:
Drug: Albuvirtide — Intravenous infusion of Albuvirtide
  Other Names: Fusion inhibitor
  Arms: Cohort 1: albuvirtide & 3BNC117; Cohort 2: albuvirtide & 3BNC117; Cohort 3: albuvirtide & 3BNC117; Cohort 4: albuvirtide & 3BNC117; Optimal Dose: albuvirtide & 3BNC117
Drug: 3BNC117 — Intravenous infusion of 3BNC117
  Other Names: Monoclonal antibody
  Arms: Cohort 1: albuvirtide & 3BNC117; Cohort 2: albuvirtide & 3BNC117; Cohort 3: albuvirtide & 3BNC117; Cohort 4: albuvirtide & 3BNC117; Optimal Dose: albuvirtide & 3BNC117
Drug: Baseline ART — Subjects continuing on baseline ART
  Other Names: ART
  Arms: Control Arm 1: Baseline ART; Control Arm 2: Baseline ART

SUMMARY:
The study is an adaptive, phase 2, multicenter, three-part study to establish the dosage, safety and antiviral activity of combination therapy with albuvirtide (ABT) and 3BNC117 as long-acting maintenance therapy in virologically suppressed subjects with HIV-1 infection.

DETAILED DESCRIPTION:
This is a three-part, multicenter study that will enroll a total of 80 eligible, HIV-1 subjects who are virologically suppressed and stable on daily oral combination antiretroviral therapy. The study will be conducted in three parts.

Part 1 and Part 2 are the dose-ranging portions of the study. In Part 1, 30 eligible subjects will be randomized in a 1:1:1 ratio to receive 16 weeks of combination treatment with albuvirtide and 3BNC117 or continue on the existing ART regimen under one of the three cohorts as follows:

* Cohort 1: albuvirtide 0.32 g and 3BNC117 2 g every 2 weeks
* Cohort 2: albuvirtide 0.32 g and 3BNC117 2 g every 4 weeks
* Control Arm 1: Subjects continuing on baseline ART

In Part 2 of the study, 20 eligible subjects will be randomized in a 1:1 ratio to receive 16 weeks of combination treatment with albuvirtide and 3BNC117 under one of the two cohorts as follows:

* Cohort 3: albuvirtide 0.32 g and 3BNC117 0.8 g every 4 weeks
* Cohort 4: albuvirtide 0.16 g and 3BNC117 0.8 g every 4 weeks

Part 3 of this study will enroll an additional 30 subjects in a 2:1 ratio to receive up to 28 weeks of combination treatment with optimal dose of albuvirtide and 3BNC117 or continue on the existing ART regimen as follows:

* Optimal Dose: albuvirtide and 3BNC11 every 2 or 4 weeks
* Control Arm 2: Subjects continuing on baseline ART All consenting patients, in Cohort 1 and 2 (Part 1) and Cohort 3 and 4 (Part 2) of the study, will be shifted from daily oral combination antiretroviral regimen to an intravenous infusion of ABT and 3BNC117. The total treatmentduration with the ABT and 3BNC117 combination regimen will be up to 16 weeks (for Part 1 and Part 2) or 28 weeks (for Part 3) with a two week overlap of the baseline oral antiretroviral regimen and the ABT-3BNC117 combination regimen at the beginning of the study treatment and at the end of the treatment phase in subjects who do not experience virologic rebound. During the two week overlap of baseline oral antiretrovirals and ABT-3BNC117 combination regimen at the beginning of the study treatment, subject will receive weekly doses of ABT and 3BNC117 as intravenous infusions. Beyond the overlap period, subjects in Cohort 1 will receive study treatments every two weeks and subjects in Cohort 2, 3, and 4 will receive study treatments every four weeks.

Study participants will be monitored for viral rebound every two weeks following initiation of ABT-3BNC117 combination and will re-initiate an oral antiretroviral regimen if virologic rebound is confirmed with plasma HIV-1 RNA levels above 200 copies/ml on two consecutive blood draws.

Pharmacokinetics of ABT and 3BNC117 will be assessed in this study.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects are required to meet all of the following criteria for enrollment into the study.

  1. HIV-1 seropositive;
  2. Males and females, age ≥18 years;
  3. Receiving oral combination antiretroviral therapy for last 24 weeks;
  4. No change in antiretroviral regimen within last 4 weeks prior to Screening Visit and in-between Screening Visit and First Treatment Visit with an exception that subjects on NNRTI-containing regimens will be allowed to switch to protease inhibitor- or integrase strand transferase inhibitor-based regimens and such change, if needed, should occur at least 4 weeks prior to cessation of oral antiretroviral therapy;
  5. Subject has two or more potential alternative antiretroviral drug options available;
  6. Plasma HIV-1 RNA <50 copies/mL at Screening Visit as determined by Human Immunodeficiency Virus 1 (HIV-1) Quantitative, RNA (Taqman® Real-Time PCR);
  7. No documented detectable viral loads (HIV-1 RNA > 50 copies/mL) within the last 24 weeks prior to Screening Visit. An exception for a recorded HIV-1 RNA "blip" (e.g., transient HIV-1 RNA <400 copies/mL) can be considered, although the preceding and following HIV-1 RNA measurements should be <50 copies/mL;
  8. CD4 cell count of >300 cells/mm3 at Screening Visit;
  9. Laboratory values at Screening:

     1. Absolute neutrophil count (ANC) ≥750/ mm3;
     2. Hemoglobin (Hb) ≥10.5 gm/dL (male) or ≥9.5 gm/dL (female);
     3. Platelets ≥75,000 /mm3;
     4. Serum alanine transaminase (SGPT/ALT) <1.25 x upper limit of normal (ULN);
     5. Serum aspartate transaminase (SGOT/AST) <1.25 x ULN;
     6. Serum total bilirubin within normal range; and
     7. Creatinine ≤1.5 x ULN.
  10. Clinically normal resting 12-lead ECG at Screening Visit or, if abnormal, considered not clinically significant by the Principal Investigator;
  11. Both male and female subjects and their partners of childbearing potential must agree to use 2 medically accepted methods of contraception (e.g., barrier contraceptives [male condom, female condom, or diaphragm with a spermicidal gel], hormonal contraceptives [implants, injectables, combination oral contraceptives, transdermal patches, or contraceptive rings], and intrauterine devices) during the course of the study (excluding women who are not of childbearing potential and men who have been sterilized or who do not have sex with women). Females of childbearing potential must have a negative serum pregnancy test at Screening visit and negative urine pregnancy test prior to receiving the first dose of study drug;
  12. Willing and able to participate in all aspects of the study, including use of intravenous medication, completion of subjective evaluations, attendance at scheduled clinic visits, and compliance with all protocol requirements as evidenced by providing written informed consent.

Note: Subjects diagnosed with either substance dependence or substance abuse or any history of a concomitant condition (e.g., medical, psychologic, or psychiatric) may be enrolled if in the opinion of site investigator these circumstances would not interfere with the subject's successful completion of the study requirements.

Exclusion Criteria:

* Potential subjects meeting any of the following criteria will be excluded from enrollment.

  1. Any active infection or malignancy requiring acute therapy;
  2. Hepatitis B infection as manifest by the presence of Hepatitis B surface antigen (HBsAg);
  3. Hepatitis C infection as manifest by positive anti-HCV antibody and positive HCV RNA assay at the time of screening;
  4. Grade 4 DAIDS laboratory abnormality;
  5. Females who are pregnant, lactating, or breastfeeding, or who plan to become pregnant during the study;
  6. Unexplained fever or clinically significant illness within 1 week prior to the first study dose;
  7. Any vaccination within 2 weeks prior to the first study dose;
  8. Subjects weighing <35kg;
  9. History of anaphylaxis to any oral or parenteral drugs;
  10. Use of any fusion inhibitors and broadly neutralizing monoclonal antibody prior to the Screening Visit;
  11. Participation in an experimental drug trial(s) within 30 days of the Screening Visit;
  12. Any known allergy or antibodies to the study drug or excipients;
  13. Treatment with any of the following:

      1. Radiation or cytotoxic chemotherapy with 30 days prior to the screening visit;
      2. Immunosuppressants or immunomodulating agents within 60 days prior to the screening visit; or
      3. Oral or parenteral corticosteroids within 30 days prior to the Screening Visit. Subjects on chronic steroid therapy > 5 mg/day will be excluded with the following exception:

         * Subjects on inhaled, nasal, or topical steroids will not be excluded.
  14. Any other clinical condition that, in the Investigator's judgment, would potentially compromise study compliance or the ability to evaluate safety/efficacy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-12-17 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with HIV-1 RNA < 50 copies/mL at the end of treatment phase in Part 3 of the study. | 28 weeks in Part 3

SECONDARY OUTCOMES:
Proportion of participants with HIV-1 RNA < 50 copies/mL at the end of treatment phase in Part 1 of the study | 16 weeks in Part 1
Proportion of participants with HIV-1 RNA < 50 copies/mL at the end of treatment phase in Part 2 of the study | 16 weeks in Part 2
Time to virologic rebound after discontinuation of baseline ART regimen | 16 weeks in Part 1 and part 2, 28 weeks in part 3
  Note: Virologic rebound is defined as two consecutive HIV-1 RNA levels of > 200 copies/ml.
Proportion of participants achieving HIV-1 RNA < 50 copies/mL after experiencing virologic rebound | 16 weeks in Part 1 and part 2, 28 weeks in part 3
Time to achieving HIV-1 RNA < 50 copies/mL after experiencing virologic rebound | 16 weeks in Part 1 and part 2, 28 weeks in part 3
Mean change in HIV-1 RNA, at each visit within the treatment phase | 16 weeks in Part 1 and part 2, 28 weeks in part 3
Mean change in CD4 cell count, at each visit within the treatment phase | 16 weeks in Part 1 and part 2, 28 weeks in part 3
Mean change in CD4:CD8 ratio, at each visit within the treatment phase | 16 weeks in Part 1 and part 2, 28 weeks in part 3
Emergence of new resistance mutations to antiretroviral drugs as evaluated by GenoSure Archive or PhenoSense GT Assay | 16 weeks in Part 1 and part 2, 28 weeks in part 3
Measurement of treatment adherence to the ABT and 3BNC117 combination regimen | 16 weeks in Part 1 and part 2, 28 weeks in part 3

CONTACTS AND LOCATIONS:
Overall Officials: Frontier clinical team, Study Director — Frontier Biotechnologies Inc.
Locations (7):
- United States (7):
  - ABT-3BNC117_201 Investigational Site, Palm Springs, California
  - ABT-3BNC117_201 Investigational Site, San Francisco, California
  - ABT-3BNC117_201 Investigational Site, Ft. Pierce, Florida
  - ABT-3BNC117_201 Investigational Site, Hialeah, Florida
  - ABT-3BNC117_201 Investigational Site, Orlando, Florida
  - ABT-3BNC117_201 Investigational Site, Atlanta, Georgia
  - ABT-3BNC117_201 Investigational Site, New York, New York

IPD SHARING:
Plan to Share IPD: No